CLINICAL TRIAL: NCT06207682
Title: An Open-Label, Phase 1 Study to Evaluate the Effect of Repeated Oral Doses of Avacopan on the Pharmacokinetics of a Single Dose of Simvastatin in Healthy Volunteers
Brief Title: Effect of Repeated Oral Doses of Avacopan on the Pharmacokinetics (PK) of a Single Dose of Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CL020_168
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: Avacopan; CCX168; Simvastatin
MeSH Terms: interventions — avacopan; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Avacopan and Simvastatin (Experimental): A single dose of 40 mg simvastatin will be given orally in the morning on Day 1 and Day 10. The Day 10 dose of simvastatin will be co-administered with the morning dose of avacopan. On Days 3 through 11, avacopan will be given orally at 30 mg BID.
  Interventions: Drug: Avacopan; Drug: Simvastatin
- Arm 2: Avacopan and Simvastatin (Experimental): A single dose of 40 mg simvastatin will be given orally in the morning on Day 1 and Day 10. The Day 10 dose of simvastatin will be co-administered with the morning dose of avacopan. On Days 3 through 11, avacopan will be given orally at 60 mg BID.
  Interventions: Drug: Avacopan; Drug: Simvastatin

INTERVENTIONS:
Drug: Avacopan — Orally via capsules
  Other Names: CCX168
Drug: Simvastatin — Orally via tablets

SUMMARY:
The primary objective of this clinical study is to evaluate the effect of repeated oral doses of avacopan (30 mg and 60 mg twice daily approximately 12 hours apart [BID]) given under fed conditions on the PK of a single dose of simvastatin (40 mg) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, 18-55 years of age, inclusive.
2. Body mass index (BMI) is 18.5 to 29.9 kg/m^2.
3. Negative result of the human immunodeficiency virus (HIV) screen, the hepatitis B screen, the hepatitis C screen, and the QuantiFERON®-TB Gold test.
4. A female participant is eligible to participate if she is of:

   1. Non-childbearing potential defined as pre-menopausal females with a documented bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy (removal of the ovaries) or hysterectomy; hysteroscopic sterilization, or post-menopausal defined as ≥12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] in the post-menopausal range is confirmatory). Documented verbal history from the participant is acceptable for all of the criteria stipulated above.
   2. Child-bearing potential and agrees to use effective contraception methods from the signing of informed consent until 120 days after the last dose of study treatment.
   3. Lactating but willing to stop breast feeding prior to the first dose of study treatment until 120 days after the last dose of study treatment.
5. Female participants must agree not to donate ova starting at Screening and for 120 days after the final study drug administration.
6. Male participants must agree to use highly effective contraception methods. This criterion must be followed from the time of the first dose of study treatment until 120 days after the last dose of study treatment.
7. Male participants must agree not to donate sperm starting from the time of the first dose of study treatment and for 120 days after the final study drug administration
8. Judged by the Investigator to be otherwise fit for the study, based on medical history, physical examination, and clinical laboratory assessments. Participants with clinical laboratory values that are outside of normal limits (other than those specified in the Exclusion Criteria) and/or with other abnormal clinical findings that are judged by the Investigator not to compromise participant participation in the study, may be entered into the study
9. Willing and able to provide written Informed Consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or have a positive serum pregnancy test at Screening or on Study Day -1 or women who desire to begin a family or breastfeed during the full length of the study.
2. Expected requirement for use of any medication (with the exception of continued use by female participants of hormonal contraceptives in accordance with a regimen that has been stable for at least the three months prior to Screening and post-menopausal females using estrogen replacement therapy) from Screening through the end of the study.
3. History within the 60 days prior to the first administration of Investigational Product (IP) of use of cannabis, tobacco and/or nicotine-containing products.
4. History of drug abuse (either illicit or prescription) within two years prior to first administration of IP.
5. History of alcohol abuse at any time in the past five years from Screening.
6. History or presence of any form of cancer within the 5 years prior to screening, with the exception of excised basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ such as cervical or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis.
7. History or presence of any medical condition or disease or laboratory abnormality which, in the opinion of the Investigator, may place the participant at unacceptable risk for study participation.
8. Donated or lost more than 50 mL of blood or blood products within 56 days prior to screening, or donated plasma within 7 days of randomization.
9. Hemoglobin less than the lower limit of normal or recent history (6 months prior to first dose) of iron deficient anemia.
10. Received a live vaccine or a vaccine for coronavirus 19 disease (COVID-19) within 4 weeks prior to Screening
11. Current or recent COVID-19 infection defined as:

    1. positive result of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-V2) test at screening or Day-1, or
    2. symptomatic COVID-19 infection within 30 days prior to Day-1, or
    3. continuing COVID-19 long haul symptomatology regardless of when the initial COVID-19 infection occurred
12. Known hypersensitivity to avacopan or inactive ingredients of the avacopan capsules (including gelatin, polyethylene glycol, or Cremophor).
13. Participated in any clinical study of an Investigational Product within 30 days or of 5 half-lives prior to randomization.
14. Participant has any evidence of hepatic disease; aspartate aminotransaminase (AST), alanine aminotransaminase (ALT), alkaline phosphatase, or bilirubin > the upper limit of normal during screening and Day -1.
15. Participant has any evidence of renal impairment, defined as estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m^2 during screening or Day-1
16. Participant's urine tested positive at Screening and/or on Study Day -1 for any of the following: opioids, opiates, amphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine, or alcohol (Breathalyzer test allowed for alcohol).
17. Use of alcohol-, caffeine-, or xanthine-containing products within 1 week prior to Day -1.
18. Participant has any evidence of gastro-intestinal disease by exam or history (not including appendectomy or hernia) which could interfere with oral absorption, digestion, or uptake. Participants with cholecystectomy should be excluded.
19. Use of any prescription medications (with the exception of hormonal contraceptives and hormonal therapy), over-the-counter nonsteroidal anti-inflammatory drugs, herbal preparations, St. John's Wort or consumption of grapefruit juice, grapefruit, or Seville oranges within 14 days before Day 1 (first dose).
20. Use of over-the-counter medications, vitamins, or supplements (including omega-3 fish oils) within 7 days before Day 1 (first dose)
21. Participants taking strong cytochrome P450 (CYP)3A4 inducers (e.g., phenytoin, fosphenytoin, rifampin, carbamazepine, St. John's Wort, nevirapine, pentobarbital, primidone, rifapentine, enzalutamide, lumacaftor, mitotane, apalutamide, quinine, rimexolone, rifaximin, rifamycin, topiramate, oxcarbazepine) or moderate CYP3A4 inducers (e.g., bosentan, efavirenz, etravirine, modafinil, dexamethasone, etravirine, nafcillin, dabrafenib, methotrexate, bexarotene, mifepristone) within 2 weeks prior to Day 1.
22. Participants taking strong CYP3A4 inhibitors (e.g., boceprevir, clarithromycin, conivaptan, grapefruit juice or grapefruit, Seville oranges, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin and voriconazole) within 2 weeks prior to Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Simvastatin | Up to Day 12
Cmax of β-hydroxy-simvastatin Acid | Up to Day 12
Area Under the Plasma Concentration-time Curve from Time 0 to the Time Point of Last Quantifiable Plasma Concentration (AUClast) of Simvastatin | Up to Day 12
AUClast of β-hydroxy-simvastatin Acid | Up to Day 12
Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUCinf) of Simvastatin | Up to Day 12
AUCinf of β-hydroxy-simvastatin Acid | Up to Day 12

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to Day 26
Cmax of Avacopan | Up to Day 12
Cmax of Avacopan Metabolite M1 | Up to Day 12
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCtau) of Avacopan | Up to Day 12
AUCtau of Avacopan Metabolite M1 | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Miao S, Bekker P, Armas D, Lor M, Han Y, Webster K, Trivedi A. Pharmacokinetic Evaluation of the CYP3A4 and CYP2C9 Drug-Drug Interaction of Avacopan in 2 Open-Label Studies in Healthy Participants. Clin Pharmacol Drug Dev. 2024 May;13(5):517-533. doi: 10.1002/cpdd.1389. Epub 2024 Feb 29. PMID 38423992